CLINICAL TRIAL: NCT05905042
Title: Follow-up of Recovery Condition in Survivors of Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Kuo-Chen Cheng, Chief, Chimei Medical Center
Other Study IDs: CMFHR10362(IRB10308-011)
Record Dates: First submitted 2018-01-24; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Hope to realize the recovery condition of ARDS survivors in Taiwan. It would be helpful not only to design the proper rehabilitation program but also to be a useful reference for the poor recovery patients to take hospice care if indicated.

DETAILED DESCRIPTION:
This study will enroll the participant met the diagnostic criteria of ARDS. The basic data, clinical manifestations, laboratory data and outcomes of participants will be recorded.

And the investigator will also follow up the pulse oximeter, peak expiratory flow rate, six-minute walk test and health-related quality of life measures with SF-36 in 3, 6 and 12 months after the participants were discharged from the ICU. Through this study, the investigator hope to realize the recovery condition of ARDS survivors in Taiwan.

It would be helpful not only to design the proper rehabilitation program but also to be a useful reference for the poor recovery patients to take hospice care if indicated.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients

Exclusion Criteria:

* NA

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
occurrence of postextubation stridor | 24 hours
  To determine whether treatment with corticosteroids decreases the incidence of postextubation airway obstruction in an adult intensive care unit.

SECONDARY OUTCOMES:
The actual tidal volume at expiration | 24 hours
  The actual tidal volume at expiration was measured before and after deflation of the endotracheal tube cuff as previously described (9). The difference in the actual tidal volume before and after cuff deflation was defined as the cuff leak volume (CLV).

IPD SHARING:
Plan to Share IPD: No